CLINICAL TRIAL: NCT00577954
Title: Multimodal Magnetic Resonance (MRI) Development in Comatose Patients for an Algorithm in the Prediction of Consciousness Recovery
Brief Title: Multimodal Resonance Imaging for Outcome Prediction on Coma Patients
Acronym: MRI-Coma
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P051061
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2008-12

CONDITIONS: Coma
Keywords: Coma; TBI; Stroke; SAH; Cerebral Anoxia; Multimodal MRI
MeSH Terms: conditions — Coma; Stroke; Hypoxia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients in a coma condition after a traumatic brain injury (250), stroke, cerebral anoxia or subarachnoid hemorrhage (150), for at least 7 days.
  Interventions: Procedure: Multimodal MRI

INTERVENTIONS:
Procedure: Multimodal MRI — Multimodal MRI

SUMMARY:
Stroke, traumatic head injury, subarachnoid hemorrhage and cerebral anoxia are main causes of a coma condition implying severe brain damage and thus, poor prognosis. Clinicians are often in need for a tool able to predict the awakening of these patients. Multimodal MRI, associating the traditional morphological sequences with spectroscopy-MRI (MRS) and the diffusion tensor imaging, could provide such a prediction.

DETAILED DESCRIPTION:
Predicting the awakening of patients in comas is one of the principal stakes of the current neurointensive care unit (neuroICU). Several studies and clinical practice suggest that the multimodal MRI, which associates the traditional morphological sequences (T1, T2*, FLAIR/T2), the spectroscopy-MRI (MRS) and the diffusion tensor imaging, is a tool allowing such a prediction. However, this strategy has not been yet validated. Additionally, currently there is no method of analysis including the 4 different sequences.

Objective: The goal of this study is to develop a composite score able to predict the awakening of coma patients following events such as a severe cranial trauma, ischemic or hemorrhagic cerebrovascular accident and cerebral anoxia. This composite score will be built from the results of the multimodal MRI (quantified indicator) in combination with clinical covariables (e.g., age of the patient, the mechanism of the accident (high versus low speed), etc.). The final score will aim to predict the outcome of patients at 1 year, evaluated by one of the following categories: favourable (Glasgow Outcome Scale (GOS 3+, 4, and 5) or unfavourable outcome (GOS 1, 2, and 3). GOS 3- score has been defined as minimally conscious state and GOS 3+ score as severe disability excluding cognitive sequelae.

MRI Analysis: The lesions present on the MRI will be quantified by a neuroradiologist and a dedicated clinical engineer from the coordination centre (Pitié-Salpêtrière Hospital) in a blinded way regarding patients' clinical data. Lesion load-indicators will be calculated on the sequences of FLAIR/T2, T2*, MRS and diffusion tensor imaging from a predefined analysis grid allowing the regional study of the lesions as well as the appreciation of their nature, their uni- or bilateral character and if bilateral, their symmetry.

Hypothesis and applicability: The multivariate analysis of morphological MRI, MRS and diffusion tensor imaging data, combined with the clinical covariables, will aim to develop a statistical algorithm, able to predict the clinical outcome of the patients. In the long term, it will be integrated into an expert system which will be the subject of a patent submission. The final objective is to provide the clinicians a diagnostic tool able to determine outcome of patients with severe cranial trauma and other neurological conditions such as stroke, subarachnoid hemorrhage and cerebral anoxia.

ELIGIBILITY:
Inclusion Criteria:

* Adult affiliated to the social security system
* Hospitalized in neuroICU and requiring artificial ventilation following a severe cranial trauma, an ischemic and/or hemorrhagic cerebrovascular accident and/or a cerebral anoxia
* In coma defined as not answering simple orders at least 7 days after the event
* Receiving an amount of sedatives and not being able to explain the coma
* Having a standardized intracranial pressure (≤ 15 mm Hg) and in absence of severe hemodynamic or respiratory failure so that the MRI does not represent any additional danger

Exclusion Criteria:

* Coma of infectious or toxic origin
* Coma explained by sedation
* MRI contraindication (pace maker, medical material not MRI compatible)
* Persistent intracranial hypertension contraindicating the setting in prolonged dorsal decubitus (ICP > 20 mm Hg during more than 10 minutes after positioning on decubitus)
* Severe hemodynamic failure
* Severe respiratory failure
* Life threatening extra-cerebral lesions
* Cranial trauma of ballistic origin
* Patient presenting a severe compromise of a major function bringing into play the vital outcome, with invalidity before the accident/event
* Former neurological pathology altering the clinical outcome of the cranial trauma
* Refusal of the family
* Patient protected by the law (under supervision or trusteeship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Traumatic brain injured patients, stroke patients, subarachnoid hemorrhage (SAH) patients and cerebral anoxia patients
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2006-10; Primary Completion 2010-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To define a quantified indicator resulting from the analysis of the multimodal MRI combined with clinical data to create a score to predict the 1 year outcome as measured by the dichotomized Glasgow Outcome Scale (extended version [GOSE]). | one year

SECONDARY OUTCOMES:
Relevance of the composite score to predict the clinical outcome at 1 year assessed by the Rankin score, the GOSE and the disability rating scale (DRS). | one year
Intra and inter-observer reproducibility study of the analysis of the various sequences. | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Pr Louis Puybasset,, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris Pitié Salpetriere
Locations (1):
- Assistance Publique Hopitaux de Paris Pitie Salpetriere, Paris, France

REFERENCES:
- [Derived] Puybasset L, Perlbarg V, Unrug J, Cassereau D, Galanaud D, Torkomian G, Battisti V, Lefort M, Velly L, Degos V, Citerio G, Bayen E, Pelegrini-Issac M; MRI-COMA Investigators CENTER-TBI MRI Participants and MRI Only Investigators. Prognostic value of global deep white matter DTI metrics for 1-year outcome prediction in ICU traumatic brain injury patients: an MRI-COMA and CENTER-TBI combined study. Intensive Care Med. 2022 Feb;48(2):201-212. doi: 10.1007/s00134-021-06583-z. Epub 2022 Dec 14. PMID 34904191
- [Derived] Simeone P, Auzias G, Lefevre J, Takerkart S, Coulon O, Lesimple B, Torkomian G, Battisti V, Jacquens A, Couret D, Naccache L, Bayen E, Bruder N, Perlbarg V, Puybasset L, Velly L. Long-term follow-up of neurodegenerative phenomenon in severe traumatic brain injury using MRI. Ann Phys Rehabil Med. 2022 Nov;65(6):101599. doi: 10.1016/j.rehab.2021.101599. Epub 2022 Feb 15. PMID 34718191
- [Derived] Velly L, Perlbarg V, Boulier T, Adam N, Delphine S, Luyt CE, Battisti V, Torkomian G, Arbelot C, Chabanne R, Jean B, Di Perri C, Laureys S, Citerio G, Vargiolu A, Rohaut B, Bruder N, Girard N, Silva S, Cottenceau V, Tourdias T, Coulon O, Riou B, Naccache L, Gupta R, Benali H, Galanaud D, Puybasset L; MRI-COMA Investigators. Use of brain diffusion tensor imaging for the prediction of long-term neurological outcomes in patients after cardiac arrest: a multicentre, international, prospective, observational, cohort study. Lancet Neurol. 2018 Apr;17(4):317-326. doi: 10.1016/S1474-4422(18)30027-9. Epub 2018 Feb 27. PMID 29500154
- [Derived] Luyt CE, Galanaud D, Perlbarg V, Vanhaudenhuyse A, Stevens RD, Gupta R, Besancenot H, Krainik A, Audibert G, Combes A, Chastre J, Benali H, Laureys S, Puybasset L; Neuro Imaging for Coma Emergence and Recovery Consortium. Diffusion tensor imaging to predict long-term outcome after cardiac arrest: a bicentric pilot study. Anesthesiology. 2012 Dec;117(6):1311-21. doi: 10.1097/ALN.0b013e318275148c. PMID 23135257